CLINICAL TRIAL: NCT03380780
Title: A Single-Center, Open-Label, Single Dose Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Emicizumab in Healthy Chinese Volunteers
Brief Title: A Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Emicizumab in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YP39308
Record Dates: First submitted 2017-12-13; First posted 2017-12-21 (Actual); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers; Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emicizumab (Experimental)
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — Participants will receive a single 1 milligram per kilogram of body weight (mg/kg) subcutaneous dose of emicizumab on Day 1.
  Other Names: RO5534262

SUMMARY:
This single-center, open-label study will evaluate the pharmacokinetics, safety, and tolerability of emicizumab following a single subcutaneous (SC) administration to healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male subjects, aged 20-45 years inclusive at the time of screening
* Chinese subjects must have Chinese parents and grandparents, all of whom were born in China
* A body mass index (BMI) between 19 and 24 kilograms per height in meters squared (kg/m^2), inclusive
* Able to participate and willing to give written informed consent and to comply with the study requirements

Exclusion Criteria:

* Any history or presence of a clinically significant disorder, or any other condition or disease which in the judgement of the investigator would place the subject at undue risk; interfere with absorption, distribution, metabolism, and excretion of emicizumab; or interfere with the ability of the subject to complete the study
* Major illness within 1 month prior to dosing, and/or any condition which could relapse during or immediately after the study
* Use of any prescribed or over-the-counter (OTC) medication or herbal medicine taken within 14 days prior to dosing or within 5 times the elimination half-life of the medication prior to dosing (whichever is longer), with some exceptions
* Any significant donation/loss of blood or plasma (greater than 450 milliliters) within the 3 months prior to dosing
* Regular smoker with consumption of more than 10 cigarettes per day or the equivalent amount of tobacco
* Participation within a clinical study with an investigational drug or device within the last 3 months prior to dosing
* Any clinically relevant history of hypersensitivity or allergic reactions, either spontaneous or following drug administration or exposure to foods or environmental agents
* Previous or concomitant thromboembolic disease such as deep vein thrombosis (DVT) or signs of thromboembolic disease, or family history of thromboembolic disorder such as serious DVT
* At high risk for thrombotic microangiopathy (e.g., have a previous medical or family history of thrombotic microangiopathy), in the investigator's judgment
* Previous or concomitant autoimmune or connective tissue disease
* History of tuberculosis or active tuberculosis with positive test result at screening
* Any other reason that, in the judgment of the investigator, would render the subject unsuitable for study participation

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Peking University Third Hospital, Beijing, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Emicizumab: Participants received a single 1 milligram per kilogram of body weight (mg/kg) subcutaneous dose of emicizumab under fasting conditions on Day 1.
Period: Overall Study
Arm/Group | Emicizumab
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Emicizumab
Description: Plasma concentrations of emicizumab were analyzed using a validated enzyme-linked immunosorbent assay (ELISA). Pharmacokinetics (PK) parameters were estimated using standard non-compartmental methods.
Time Frame: Predose on Day 1 and postdose on Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: The pharmacokinetics (PK) analysis population included all enrolled participants; participants were planned to be excluded if they deviated significantly from the protocol or if data was unavailable or incomplete which may influence the PK analysis.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (μg/mL)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
microgram per milliliter (μg/mL) | 7.11 (1.77)

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) Between Time Zero Extrapolated to Infinity (AUC0-inf) of Emicizumab
Description: as for outcome 1
Time Frame: Predose on Day 1 and postdose on Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
μg*day/mL | 287 (74.2)

3. Secondary Outcome: AUC Between Time Zero and the Time of Last Quantifiable Concentration (AUC0-last) of Emicizumab
Description: as for outcome 1
Time Frame: Predose on Day 1 and postdose on Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
μg*day/mL | 268 (63.7)

4. Secondary Outcome: Time to Cmax (Tmax) of Emicizumab
Description: as for outcome 1
Time Frame: Predose on Day 1 and postdose on Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 1
Measure: Median (Full Range); unit: day
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
day | 7.0 [3.0 to 15.0]

5. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Emicizumab
Description: as for outcome 1
Time Frame: Predose on Day 1 and postdose on Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
day | 26.7 (4.25)

6. Secondary Outcome: Apparent Clearance (CL/F) of Emicizumab
Description: as for outcome 1
Time Frame: Predose on Day 1 and postdose on Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliter per day (mL/day)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
milliliter per day (mL/day) | 235 (88)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Emicizumab
Description: as for outcome 1
Time Frame: Predose on Day 1 and postdose on Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
mL | 8870 (2950)

8. Secondary Outcome: Mean Residence Time (MRT) of Emicizumab
Description: as for outcome 1
Time Frame: Predose on Day 1 and postdose on Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
day | 40.26 (6.34)

9. Secondary Outcome: Number of Participants With Adverse Events by Highest World Health Organization (WHO) Toxicity Grade
Description: The WHO Toxicity Grading Scale was used for assessing adverse event severity. Any adverse event not specifically listed in the WHO Toxicity Grading Scale was assessed according to the following levels of severity: Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe; and Grade 4 is life-threatening. Investigator text for adverse events were encoded using the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. After informed consent had been obtained but prior to initiation of study drug, only serious adverse events (SAEs) caused by a protocol-mandated intervention were to have been reported. After initiation of study drug, all adverse events, regardless of relationship to study drug, were to have been reported until the participant completed his last study visit. After this period, any SAEs believed to be related to prior study drug treatment were to be reported.
Time Frame: From screening to study completion (20 weeks)
Population: The safety analysis population included all participants who had received any amount of study medication, whether prematurely withdrawn from the study or not, and with at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
Participants
  Any Adverse Event - Any Grade | 14
  Any Adverse Event - Grade 1 | 7
  Any Adverse Event - Grade 2 | 7
  Any Adverse Event - Grade 3 | 0
  Any Adverse Event - Grade 4 | 0
  Leukopenia - Grade 1 | 1
  Diarrhoea - Grade 1 | 1
  Flatulence - Grade 1 | 1
  Mouth ulceration - Grade 2 | 1
  Toothache - Grade 1 | 1
  Conjunctivitis - Grade 2 | 1
  Gastroenteritis - Grade 2 | 1
  Pericoronitis - Grade 1 | 1
  Upper respiratory tract infection - Grade 1 | 3
  Upper respiratory tract infection - Grade 2 | 1
  Injury - Grade 2 | 1
  Road traffic accident - Grade 2 | 1
  Blood bilirubin increased - Grade 1 | 1
  Blood creatinine phosphokinase increased - Grade 1 | 4
  Blood triglycerides increased - Grade 1 | 1
  Blood uric acid increased - Grade 1 | 1
  C-reactive protein increased - Grade 1 | 2
  White blood cell count decreased - Grade 1 | 1
  White blood cell count increased - Grade 1 | 1
  Hypertriglyceridaemia - Grade 1 | 1
  Hypokalaemia - Grade 2 | 1
  Cough - Grade 1 | 1
  Dry throat - Grade 1 | 1
  Nasal congestion - Grade 1 | 1
  Nasal obstruction - Grade 2 | 1
  Oropharyngeal pain - Grade 1 | 3
  Rash - Grade 1 | 1

10. Secondary Outcome: Number of Participants Testing Negative or Positive for the Presence of Anti-Drug Antibodies (ADA) Against Emicizumab by Timepoint and for the Overall Study
Description: Participants were considered to be 'ADA Negative (Treatment Unaffected)' if baseline and all post-baseline samples were negative, or if they were ADA positive at baseline but did not have any post-baseline samples with a titer that was at least 4-fold greater than the titer of the baseline sample. 'Total ADA Positive' is the sum of all participants who tested positive for ADA in the 2 following categories: 'ADA Positive (Treatment Induced)', those who were ADA negative at baseline and tested positive for ADA following study drug administration; and 'ADA Positive (Treatment Boosted)', those who were pre-dose ADA positive and had post-baseline samples with a titer that was at least 4-fold greater compared to the baseline measurement.
Time Frame: Predose at Baseline (Day 1) and postdose on Days 57 and 113
Population: Includes participants with at least one predose and one postdose anti-drug antibody (ADA) assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
Participants
  Baseline - ADA Positive | 0
  Baseline - ADA Negative | 16
  Day 57 - ADA Positive | 0
  Day 57 - ADA Negative | 16
  Day 113 - ADA Positive | 1
  Day 113 - ADA Negative | 15
  Overall - ADA Negative (Treatment Unaffected) | 15
  Overall - Total ADA Positive (Induced + Boosted) | 1
  Overall - ADA Positive (Treatment Induced) | 1
  Overall - ADA Positive (Treatment Boosted) | 0

11. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: The number of participants with a laboratory abnormality during treatment (numerator) is reported among the 'number analyzed' in the table below (denominator), which represents the number of participants without that abnormality at baseline (last observation prior to initiation of study drug). Note that samples from all participants were analyzed for each laboratory parameter. Values falling above or below the Roche predefined standard reference range were laboratory abnormalities labelled accordingly as 'high' or 'low'. Not every laboratory abnormality qualified as an adverse event; only if it was accompanied by clinical symptoms, resulted in a change in study treatment or in a medical intervention, or was clinically significant in the investigator's judgment. SGOT/AST = serum glutamic-oxaloacetic transaminase/aspartate transaminase; SGPT/ALT = serum glutamic-pyruvic transaminase/alanine transaminase
Time Frame: Baseline and Days 2, 4, 8, 11, 15, 29, 43, 57, 71, 85, and 113
Population: Safety analysis population. The number analyzed in the table below represents the number of participants without the specified laboratory abnormality at baseline. Samples from all participants were analyzed for each laboratory parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
Participants
  Albumin - Low | 1
  Alkaline Phosphatase - High | 2
  SGPT/ALT - Low | 2
  SGOT/AST - Low: number analyzed (Participants) | 12
  SGOT/AST - Low | 5
  Blood Urea Nitrogen - Low: number analyzed (Participants) | 15
  Blood Urea Nitrogen - Low | 1
  Blood Urea Nitrogen - High | 1
  Chloride - Low | 2
  Cholesterol - Low: number analyzed (Participants) | 7
  Cholesterol - Low | 5
  Cholesterol - High | 1
  Creatine Kinase - High: number analyzed (Participants) | 14
  Creatine Kinase - High | 3
  C-Reactive Protein - High | 6
  Lactate Dehydrogenase - Low: number analyzed (Participants) | 15
  Lactate Dehydrogenase - Low | 2
  Potassium - Low | 1
  Sodium - Low | 6
  Bilirubin - High: number analyzed (Participants) | 14
  Bilirubin - High | 2
  Protein, Total - Low: number analyzed (Participants) | 15
  Protein, Total - Low | 3
  Triglycerides (Fasting) - High | 6
  Uric Acid - Low | 2
  Uric Acid - High | 4
  Fibrinogen - Low: number analyzed (Participants) | 14
  Fibrinogen - Low | 2
  Activated Partial Thromboplastin Time - Low | 13
  Basophils, Absolute Count - High: number analyzed (Participants) | 15
  Basophils, Absolute Count - High | 4
  Eosinophils, Absolute Count - Low | 1
  Eosinophils, Absolute Count - High | 2
  Hematocrit - Low | 3
  Hemoglobin - High | 1
  Lymphocytes, Absolute Count - Low: number analyzed (Participants) | 15
  Lymphocytes, Absolute Count - Low | 4
  Lymphocytes, Absolute Count - High: number analyzed (Participants) | 15
  Lymphocytes, Absolute Count - High | 1
  Erythrocyte Mean Corpuscular Hemoglobin (HGB)-High: number analyzed (Participants) | 15
  Erythrocyte Mean Corpuscular Hemoglobin (HGB)-High | 1
  Erythro. Mean Corpuscular HGB Concentration - High: number analyzed (Participants) | 14
  Erythro. Mean Corpuscular HGB Concentration - High | 8
  Monocytes, Absolute Count - High | 2
  Neutrophils, Total, Absolute Count - Low | 2
  Neutrophils, Total, Absolute Count - High | 2
  Platelet - High | 1
  Red Blood Cell Count - Low | 3
  White Blood Cell Count - Low | 2
  Urine pH - High: number analyzed (Participants) | 12
  Urine pH - High | 9
  Urine Specific Gravity - Low: number analyzed (Participants) | 9
  Urine Specific Gravity - Low | 6
  Urine Specific Gravity - High: number analyzed (Participants) | 13
  Urine Specific Gravity - High | 9

12. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Albumin Concentration
Description: Blood samples were collected from participants at the indicated timepoints for evaluation of clinical chemistry parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: gram per Liter (g/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
gram per Liter (g/L)
  Baseline (BL) - Value at Visit | 45.43 (1.834)
  Change From BL at Day 2 | -0.43 (2.391)
  Change From BL at Day 4 | 1.03 (2.016)
  Change From BL at Day 8 | 0.29 (2.095)
  Change From BL at Day 15 | 0.08 (1.928)
  Change From BL at Day 29 | -0.18 (1.602)
  Change From BL at Day 43 | -0.41 (1.242)
  Change From BL at Day 57 | -1.24 (2.298)
  Change From BL at Day 71 | -0.58 (1.983)
  Change From BL at Day 85 | -1.56 (2.308)
  Change From BL at Day 113 | -0.26 (1.732)
  Post-BL Minimum Change From BL | -2.87 (1.967)
  Post-BL Maximum Change From BL | 1.98 (1.521)

13. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Alkaline Phosphatase Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: unit per Liter (U/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
unit per Liter (U/L)
  Baseline (BL) - Value at Visit | 85.38 (19.500)
  Change From BL at Day 2 | 0.50 (6.792)
  Change From BL at Day 4 | 2.50 (6.542)
  Change From BL at Day 8 | 1.06 (5.813)
  Change From BL at Day 15 | 2.38 (9.150)
  Change From BL at Day 29 | 1.44 (8.959)
  Change From BL at Day 43 | 0.56 (8.756)
  Change From BL at Day 57 | -3.69 (9.918)
  Change From BL at Day 71 | -0.94 (11.198)
  Change From BL at Day 85 | -4.50 (7.589)
  Change From BL at Day 113 | -0.38 (11.684)
  Post-BL Minimum Change From BL | -9.81 (7.556)
  Post-BL Maximum Change From BL | 9.94 (7.398)

14. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Bilirubin Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: micromole per Liter (μmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
micromole per Liter (μmol/L)
  Baseline (BL) - Value at Visit | 13.83 (7.556)
  Change From BL at Day 2 | 0.82 (2.921)
  Change From BL at Day 4 | -0.42 (4.470)
  Change From BL at Day 8 | -1.10 (3.713)
  Change From BL at Day 15 | -0.61 (5.909)
  Change From BL at Day 29 | -0.56 (4.688)
  Change From BL at Day 43 | -0.25 (3.709)
  Change From BL at Day 57 | -0.96 (4.034)
  Change From BL at Day 71 | 1.67 (7.467)
  Change From BL at Day 85 | 0.54 (3.861)
  Change From BL at Day 113 | -0.12 (5.570)
  Post-BL Minimum Change From BL | -3.94 (4.749)
  Post-BL Maximum Change From BL | 5.54 (5.909)

15. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Fasting Blood Glucose Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millimole per Liter (mmol/L)
  Baseline (BL) - Value at Visit | 5.03 (0.425)
  Change From BL at Day 2 | -0.33 (0.384)
  Change From BL at Day 4 | -0.22 (0.500)
  Change From BL at Day 8 | -0.16 (0.441)
  Change From BL at Day 15 | -0.27 (0.382)
  Change From BL at Day 29 | -0.08 (0.364)
  Change From BL at Day 43 | -0.08 (0.435)
  Change From BL at Day 57 | -0.22 (0.515)
  Change From BL at Day 71 | -0.20 (0.322)
  Change From BL at Day 85 | -0.25 (0.346)
  Change From BL at Day 113 | -0.21 (0.470)
  Post-BL Minimum Change From BL | -0.64 (0.388)
  Post-BL Maximum Change From BL | 0.24 (0.386)

16. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Blood Urea Nitrogen Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millimole per Liter (mmol/L)
  Baseline (BL) - Value at Visit | 4.46 (0.848)
  Change From BL at Day 2 | -0.58 (0.877)
  Change From BL at Day 4 | -0.73 (0.649)
  Change From BL at Day 8 | 0.26 (1.074)
  Change From BL at Day 15 | 0.43 (1.543)
  Change From BL at Day 29 | 0.43 (1.071)
  Change From BL at Day 43 | 0.38 (0.959)
  Change From BL at Day 57 | 0.39 (0.874)
  Change From BL at Day 71 | 0.36 (0.958)
  Change From BL at Day 85 | 0.16 (0.888)
  Change From BL at Day 113 | 0.13 (0.573)
  Post-BL Minimum Change From BL | -1.07 (0.587)
  Post-BL Maximum Change From BL | 1.42 (0.970)

17. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: C-Reactive Protein Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milligram per Liter (mg/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
milligram per Liter (mg/L)
  Baseline (BL) - Value at Visit | 0.50 (0.568)
  Change From BL at Day 2 | 0.23 (0.456)
  Change From BL at Day 4 | 0.11 (0.477)
  Change From BL at Day 8 | 0.54 (1.721)
  Change From BL at Day 15 | 0.75 (1.197)
  Change From BL at Day 29 | 1.01 (1.289)
  Change From BL at Day 43 | 0.60 (1.849)
  Change From BL at Day 57 | 0.27 (0.827)
  Change From BL at Day 71 | 0.13 (0.410)
  Change From BL at Day 85 | 0.12 (0.595)
  Change From BL at Day 113 | 1.24 (3.517)
  Post-BL Minimum Change From BL | -0.20 (0.397)
  Post-BL Maximum Change From BL | 3.14 (3.641)

18. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Chloride Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millimole per Liter (mmol/L)
  Baseline (BL) - Value at Visit | 104.69 (1.957)
  Change From BL at Day 2 | -0.69 (2.549)
  Change From BL at Day 4 | -0.63 (2.363)
  Change From BL at Day 8 | 0.13 (2.579)
  Change From BL at Day 15 | 0.06 (2.175)
  Change From BL at Day 29 | -1.56 (2.279)
  Change From BL at Day 43 | -0.06 (1.731)
  Change From BL at Day 57 | 0.75 (2.769)
  Change From BL at Day 71 | -0.50 (2.757)
  Change From BL at Day 85 | 0.13 (2.630)
  Change From BL at Day 113 | -0.13 (2.217)
  Post-BL Minimum Change From BL | -2.94 (2.016)
  Post-BL Maximum Change From BL | 2.31 (2.120)

19. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Cholesterol Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millimole per Liter (mmol/L)
  Baseline (BL) - Value at Visit | 3.88 (1.103)
  Change From BL at Day 2 | 0.02 (0.393)
  Change From BL at Day 4 | 0.07 (0.439)
  Change From BL at Day 8 | -0.03 (0.383)
  Change From BL at Day 15 | -0.04 (0.451)
  Change From BL at Day 29 | 0.03 (0.372)
  Change From BL at Day 43 | -0.06 (0.441)
  Change From BL at Day 57 | -0.04 (0.459)
  Change From BL at Day 71 | -0.01 (0.466)
  Change From BL at Day 85 | -0.13 (0.515)
  Change From BL at Day 113 | 0.01 (0.394)
  Post-BL Minimum Change From BL | -0.47 (0.468)
  Post-BL Maximum Change From BL | 0.47 (0.222)

20. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Creatine Kinase Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: unit per Liter (U/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
unit per Liter (U/L)
  Baseline (BL) - Value at Visit | 121.63 (81.915)
  Change From BL at Day 2 | -41.13 (54.760)
  Change From BL at Day 4 | -25.81 (107.494)
  Change From BL at Day 8 | -22.19 (54.034)
  Change From BL at Day 15 | -0.94 (39.834)
  Change From BL at Day 29 | 8.50 (122.645)
  Change From BL at Day 43 | -21.00 (53.551)
  Change From BL at Day 57 | 8.00 (152.217)
  Change From BL at Day 71 | -19.63 (51.798)
  Change From BL at Day 85 | -20.00 (77.283)
  Change From BL at Day 113 | -18.81 (71.191)
  Post-BL Minimum Change From BL | -52.38 (72.902)
  Post-BL Maximum Change From BL | 92.50 (155.002)

21. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Creatinine Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: micromole per Liter (μmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
micromole per Liter (μmol/L)
  Baseline (BL) - Value at Visit | 83.19 (7.195)
  Change From BL at Day 2 | -0.56 (7.071)
  Change From BL at Day 4 | -0.31 (5.147)
  Change From BL at Day 8 | -1.25 (4.919)
  Change From BL at Day 15 | -2.00 (9.452)
  Change From BL at Day 29 | -3.69 (4.672)
  Change From BL at Day 43 | -2.06 (5.434)
  Change From BL at Day 57 | -2.38 (5.488)
  Change From BL at Day 71 | -1.06 (7.344)
  Change From BL at Day 85 | -1.50 (4.662)
  Change From BL at Day 113 | -0.19 (6.327)
  Post-BL Minimum Change From BL | -9.25 (5.170)
  Post-BL Maximum Change From BL | 6.13 (6.109)

22. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Direct Bilirubin Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: micromole per Liter (μmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
micromole per Liter (μmol/L)
  Baseline (BL) - Value at Visit | 1.63 (0.567)
  Change From BL at Day 2 | 0.56 (0.395)
  Change From BL at Day 4 | 0.29 (0.452)
  Change From BL at Day 8 | 0.00 (0.327)
  Change From BL at Day 15 | -0.07 (0.521)
  Change From BL at Day 29 | 0.12 (0.548)
  Change From BL at Day 43 | 0.12 (0.308)
  Change From BL at Day 57 | -0.03 (0.342)
  Change From BL at Day 71 | 0.23 (0.509)
  Change From BL at Day 85 | 0.17 (0.515)
  Change From BL at Day 113 | 0.07 (0.480)
  Post-BL Minimum Change From BL | -0.39 (0.396)
  Post-BL Maximum Change From BL | 0.78 (0.448)

23. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Gamma Glutamyl Transferase Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: unit per Liter (U/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
unit per Liter (U/L)
  Baseline (BL) - Value at Visit | 19.94 (10.951)
  Change From BL at Day 2 | -0.50 (1.862)
  Change From BL at Day 4 | 0.13 (1.996)
  Change From BL at Day 8 | 0.19 (3.016)
  Change From BL at Day 15 | -0.13 (10.379)
  Change From BL at Day 29 | -0.13 (3.202)
  Change From BL at Day 43 | -0.13 (3.845)
  Change From BL at Day 57 | -0.25 (4.712)
  Change From BL at Day 71 | 0.13 (5.353)
  Change From BL at Day 85 | -0.69 (3.790)
  Change From BL at Day 113 | 1.75 (5.756)
  Post-BL Minimum Change From BL | -4.81 (7.901)
  Post-BL Maximum Change From BL | 5.94 (6.319)

24. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Lactate Dehydrogenase Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: unit per Liter (U/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
unit per Liter (U/L)
  Baseline (BL) - Value at Visit | 153.75 (22.228)
  Change From BL at Day 2 | -10.13 (13.495)
  Change From BL at Day 4 | -0.19 (15.246)
  Change From BL at Day 8 | 3.19 (11.053)
  Change From BL at Day 15 | 3.19 (17.505)
  Change From BL at Day 29 | 6.56 (17.397)
  Change From BL at Day 43 | 2.38 (11.730)
  Change From BL at Day 57 | 1.69 (11.247)
  Change From BL at Day 71 | 0.19 (15.003)
  Change From BL at Day 85 | 2.63 (16.536)
  Change From BL at Day 113 | -0.38 (16.141)
  Post-BL Minimum Change From BL | -16.06 (11.168)
  Post-BL Maximum Change From BL | 22.00 (13.765)

25. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Potassium Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millimole per Liter (mmol/L)
  Baseline (BL) - Value at Visit | 4.27 (0.351)
  Change From BL at Day 2 | 0.11 (0.401)
  Change From BL at Day 4 | -0.03 (0.307)
  Change From BL at Day 8 | 0.12 (0.316)
  Change From BL at Day 15 | -0.02 (0.351)
  Change From BL at Day 29 | -0.05 (0.337)
  Change From BL at Day 43 | 0.06 (0.366)
  Change From BL at Day 57 | 0.05 (0.507)
  Change From BL at Day 71 | -0.04 (0.320)
  Change From BL at Day 85 | -0.19 (0.317)
  Change From BL at Day 113 | -0.05 (0.371)
  Post-BL Minimum Change From BL | -0.47 (0.311)
  Post-BL Maximum Change From BL | 0.45 (0.248)

26. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Total Protein Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: gram per Liter (g/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
gram per Liter (g/L)
  Baseline (BL) - Value at Visit | 70.55 (3.485)
  Change From BL at Day 2 | -0.18 (4.502)
  Change From BL at Day 4 | 2.69 (3.711)
  Change From BL at Day 8 | 1.36 (3.458)
  Change From BL at Day 15 | 0.81 (3.837)
  Change From BL at Day 29 | 1.03 (2.632)
  Change From BL at Day 43 | -0.03 (2.452)
  Change From BL at Day 57 | -1.41 (3.502)
  Change From BL at Day 71 | 0.17 (3.720)
  Change From BL at Day 85 | -1.13 (4.063)
  Change From BL at Day 113 | 0.71 (3.779)
  Post-BL Minimum Change From BL | -3.95 (3.488)
  Post-BL Maximum Change From BL | 4.54 (2.451)

27. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: SGOT/AST Concentration
Description: Blood samples were collected from participants at the indicated timepoints for evaluation of clinical chemistry parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last sample prior to initiation of study drug. SGOT/AST = serum glutamic-oxaloacetic transaminase/aspartate transaminase
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: unit per Liter (U/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
unit per Liter (U/L)
  Baseline (BL) - Value at Visit | 16.63 (2.918)
  Change From BL at Day 2 | -0.81 (2.007)
  Change From BL at Day 4 | 1.13 (2.941)
  Change From BL at Day 8 | 0.69 (3.240)
  Change From BL at Day 15 | 0.19 (3.728)
  Change From BL at Day 29 | 1.13 (3.304)
  Change From BL at Day 43 | -0.25 (1.770)
  Change From BL at Day 57 | 0.69 (3.219)
  Change From BL at Day 71 | -0.31 (2.798)
  Change From BL at Day 85 | -0.63 (2.778)
  Change From BL at Day 113 | -0.19 (3.920)
  Post-BL Minimum Change From BL | -2.94 (2.594)
  Post-BL Maximum Change From BL | 4.75 (3.416)

28. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: SGPT/ALT Concentration
Description: Blood samples were collected from participants at the indicated timepoints for evaluation of clinical chemistry parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last sample prior to initiation of study drug. SGPT/ALT = serum glutamic-pyruvic transaminase/alanine transaminase
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: unit per Liter (U/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
unit per Liter (U/L)
  Baseline (BL) - Value at Visit | 15.63 (6.449)
  Change From BL at Day 2 | -0.31 (2.798)
  Change From BL at Day 4 | 2.19 (5.419)
  Change From BL at Day 8 | 2.19 (3.953)
  Change From BL at Day 15 | -0.13 (7.702)
  Change From BL at Day 29 | 0.25 (6.340)
  Change From BL at Day 43 | -1.69 (5.199)
  Change From BL at Day 57 | -1.13 (6.490)
  Change From BL at Day 71 | -0.50 (6.408)
  Change From BL at Day 85 | -1.13 (5.560)
  Change From BL at Day 113 | -0.63 (7.571)
  Post-BL Minimum Change From BL | -5.13 (6.206)
  Post-BL Maximum Change From BL | 8.25 (6.943)

29. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Sodium Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millimole per Liter (mmol/L)
  Baseline (BL) - Value at Visit | 140.56 (1.590)
  Change From BL at Day 2 | -0.44 (1.931)
  Change From BL at Day 4 | -0.44 (1.931)
  Change From BL at Day 8 | -0.06 (2.594)
  Change From BL at Day 15 | 0.25 (1.612)
  Change From BL at Day 29 | -1.75 (2.671)
  Change From BL at Day 43 | -0.13 (2.062)
  Change From BL at Day 57 | 0.06 (2.932)
  Change From BL at Day 71 | -1.25 (3.130)
  Change From BL at Day 85 | -0.38 (2.705)
  Change From BL at Day 113 | -0.13 (1.893)
  Post-BL Minimum Change From BL | -3.38 (2.391)
  Post-BL Maximum Change From BL | 2.31 (1.922)

30. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Fasting Triglycerides Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millimole per Liter (mmol/L)
  Baseline (BL) - Value at Visit | 0.98 (0.446)
  Change From BL at Day 2 | 0.37 (0.377)
  Change From BL at Day 4 | 0.57 (0.517)
  Change From BL at Day 8 | 0.03 (0.350)
  Change From BL at Day 15 | 0.22 (0.497)
  Change From BL at Day 29 | 0.15 (0.382)
  Change From BL at Day 43 | 0.17 (0.278)
  Change From BL at Day 57 | 0.27 (0.726)
  Change From BL at Day 71 | 0.14 (0.314)
  Change From BL at Day 85 | 0.28 (0.395)
  Change From BL at Day 113 | 0.33 (0.429)
  Post-BL Minimum Change From BL | -0.19 (0.318)
  Post-BL Maximum Change From BL | 1.02 (0.490)

31. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Test Results by Timepoint: Uric Acid Concentration
Description: as for outcome 12
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: micromole per Liter (μmol/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
micromole per Liter (μmol/L)
  Baseline (BL) - Value at Visit | 323.44 (52.081)
  Change From BL at Day 2 | 21.38 (28.329)
  Change From BL at Day 4 | -15.06 (38.979)
  Change From BL at Day 8 | -2.88 (35.955)
  Change From BL at Day 15 | 2.44 (49.536)
  Change From BL at Day 29 | 2.31 (32.946)
  Change From BL at Day 43 | 9.63 (45.045)
  Change From BL at Day 57 | 9.38 (53.799)
  Change From BL at Day 71 | 33.81 (84.440)
  Change From BL at Day 85 | 19.25 (50.464)
  Change From BL at Day 113 | 34.56 (62.406)
  Post-BL Minimum Change From BL | -39.94 (25.870)
  Post-BL Maximum Change From BL | 79.25 (62.143)

32. Secondary Outcome: Change From Baseline in Coagulation Laboratory Test Results by Timepoint: Activated Partial Thromboplastin Time
Description: Blood samples were collected from participants at the indicated timepoints for evaluation of coagulation parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 11, 29, 57, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
second
  Baseline (BL) - Value at Visit | 31.63 (2.111)
  Change From BL at Day 2 | -2.79 (1.626)
  Change From BL at Day 11 | -4.82 (1.466)
  Change From BL at Day 29 | -3.63 (1.643)
  Change From BL at Day 57 | -2.14 (1.177)
  Change From BL at Day 113 | -0.70 (1.517)
  Post-BL Minimum Change From BL | -4.83 (1.482)
  Post-BL Maximum Change From BL | -0.56 (1.463)

33. Secondary Outcome: Change From Baseline in Coagulation Laboratory Test Results by Timepoint: Fibrinogen Concentration
Description: as for outcome 32
Time Frame: Baseline and Days 2, 11, 29, 57 and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: gram per Liter (g/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
gram per Liter (g/L)
  Baseline (BL) - Value at Visit | 2.43 (0.410)
  Change From BL at Day 2 | 0.18 (0.281)
  Change From BL at Day 11 | 0.28 (0.314)
  Change From BL at Day 29 | 0.11 (0.312)
  Change From BL at Day 57 | 0.05 (0.285)
  Change From BL at Day 113 | 0.07 (0.438)
  Post-BL Minimum Change From BL | -0.17 (0.222)
  Post-BL Maximum Change From BL | 0.53 (0.290)

34. Secondary Outcome: Change From Baseline in Coagulation Laboratory Test Results by Timepoint: Prothrombin Time
Description: as for outcome 32
Time Frame: Baseline and Days 2, 11, 29, 57 and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
second
  Baseline (BL) - Value at Visit | 11.33 (0.685)
  Change From BL at Day 2 | 0.00 (0.502)
  Change From BL at Day 11 | -0.09 (0.463)
  Change From BL at Day 29 | -0.18 (0.455)
  Change From BL at Day 57 | -0.18 (0.508)
  Change From BL at Day 113 | -0.17 (0.632)
  Post-BL Minimum Change From BL | -0.58 (0.457)
  Post-BL Maximum Change From BL | 0.37 (0.480)

35. Secondary Outcome: Change From Baseline in Coagulation Laboratory Test Results by Timepoint: Prothrombin Time/International Normalized Ratio (INR)
Description: The INR is a standardized measure of the prothrombin time. Blood samples were collected from participants at the indicated timepoints for evaluation of coagulation parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 11, 29, 57 and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: INR of prothrombin time (sec/sec)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
INR of prothrombin time (sec/sec)
  Baseline (BL) - Value at Visit | 1.06 (0.062)
  Change From BL at Day 2 | 0.00 (0.044)
  Change From BL at Day 11 | -0.01 (0.043)
  Change From BL at Day 29 | -0.02 (0.042)
  Change From BL at Day 57 | -0.02 (0.046)
  Change From BL at Day 113 | -0.02 (0.057)
  Post-BL Minimum Change From BL | -0.05 (0.042)
  Post-BL Maximum Change From BL | 0.03 (0.043)

36. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Basophils, Absolute Count
Description: Blood samples were collected from participants at the indicated timepoints for evaluation of hematology parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: *10^9 cells per Liter
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
*10^9 cells per Liter
  Baseline (BL) - Value at Visit | 0.02 (0.018)
  Change From BL at Day 2 | 0.00 (0.013)
  Change From BL at Day 4 | 0.01 (0.018)
  Change From BL at Day 8 | 0.01 (0.029)
  Change From BL at Day 15 | 0.01 (0.022)
  Change From BL at Day 29 | 0.01 (0.014)
  Change From BL at Day 43 | 0.01 (0.023)
  Change From BL at Day 57 | 0.01 (0.016)
  Change From BL at Day 71 | 0.01 (0.022)
  Change From BL at Day 85 | 0.00 (0.021)
  Change From BL at Day 113 | 0.01 (0.019)
  Post-BL Minimum Change From BL | -0.01 (0.016)
  Post-BL Maximum Change From BL | 0.03 (0.021)

37. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Eosinophils, Absolute Count
Description: as for outcome 36
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: *10^9 cells per Liter
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
*10^9 cells per Liter
  Baseline (BL) - Value at Visit | 0.14 (0.122)
  Change From BL at Day 2 | 0.02 (0.063)
  Change From BL at Day 4 | 0.01 (0.066)
  Change From BL at Day 8 | 0.00 (0.066)
  Change From BL at Day 15 | -0.01 (0.074)
  Change From BL at Day 29 | -0.01 (0.055)
  Change From BL at Day 43 | 0.00 (0.101)
  Change From BL at Day 57 | -0.02 (0.055)
  Change From BL at Day 71 | 0.01 (0.102)
  Change From BL at Day 85 | -0.02 (0.063)
  Change From BL at Day 113 | 0.02 (0.121)
  Post-BL Minimum Change From BL | -0.06 (0.080)
  Post-BL Maximum Change From BL | 0.07 (0.085)

38. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Erythrocyte Mean Corpuscular Hemoglobin
Description: Erythrocyte mean corpuscular hemoglobin (MCH) is a measure of the average amount of hemoglobin per red blood cell. Blood samples were collected from participants at the indicated timepoints for evaluation of hematology parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: picogram per cell
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
picogram per cell
  Baseline (BL) - Value at Visit | 30.84 (1.815)
  Change From BL at Day 2 | 0.23 (0.467)
  Change From BL at Day 4 | 0.09 (0.473)
  Change From BL at Day 8 | 0.26 (0.594)
  Change From BL at Day 15 | -0.12 (0.472)
  Change From BL at Day 29 | 0.04 (0.507)
  Change From BL at Day 43 | 0.48 (0.493)
  Change From BL at Day 57 | 0.28 (0.567)
  Change From BL at Day 71 | 0.40 (0.625)
  Change From BL at Day 85 | 0.39 (0.738)
  Change From BL at Day 113 | 0.51 (0.933)
  Post-BL Minimum Change From BL | -0.40 (0.412)
  Post-BL Maximum Change From BL | 1.24 (0.730)

39. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Erythrocyte Mean Corpuscular Volume
Description: Erythrocyte mean corpuscular volume is a measure of the average volume of a red blood cell. Blood samples were collected from participants at the indicated timepoints for evaluation of hematology parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
femtoliter (fL)
  Baseline (BL) - Value at Visit | 89.79 (3.689)
  Change From BL at Day 2 | -0.14 (1.172)
  Change From BL at Day 4 | 0.01 (0.954)
  Change From BL at Day 8 | 0.21 (1.138)
  Change From BL at Day 15 | 0.88 (1.036)
  Change From BL at Day 29 | -0.08 (0.849)
  Change From BL at Day 43 | 1.41 (1.670)
  Change From BL at Day 57 | 1.04 (1.488)
  Change From BL at Day 71 | 0.85 (1.498)
  Change From BL at Day 85 | 0.86 (1.656)
  Change From BL at Day 113 | 0.62 (1.775)
  Post-BL Minimum Change From BL | -1.17 (0.899)
  Post-BL Maximum Change From BL | 2.34 (1.138)

40. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Erythrocyte Mean Corpuscular Hemoglobin Concentration
Description: Erythrocyte mean corpuscular hemoglobin concentration (MCHC) is a measure of the average concentration of hemoglobin per red blood cell. Blood samples were collected from participants at the indicated timepoints for evaluation of hematology parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: gram per Liter (g/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
gram per Liter (g/L)
  Baseline (BL) - Value at Visit | 343.25 (8.790)
  Change From BL at Day 2 | 3.13 (6.438)
  Change From BL at Day 4 | 1.00 (7.239)
  Change From BL at Day 8 | 2.31 (5.606)
  Change From BL at Day 15 | -4.56 (6.562)
  Change From BL at Day 29 | 0.69 (6.019)
  Change From BL at Day 43 | 0.13 (8.853)
  Change From BL at Day 57 | -0.75 (8.798)
  Change From BL at Day 71 | 1.25 (6.372)
  Change From BL at Day 85 | 1.13 (8.277)
  Change From BL at Day 113 | 3.25 (8.004)
  Post-BL Minimum Change From BL | -9.00 (6.143)
  Post-BL Maximum Change From BL | 10.56 (6.099)

41. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Hematocrit (as a Fraction of 1)
Description: Hematocrit is a measure of the ratio of red blood cells (RBCs) in the blood by volume. Blood samples were collected from participants at the indicated timepoints for evaluation of hematology parameters. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio of RBCs in blood (L/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
ratio of RBCs in blood (L/L)
  Baseline (BL) - Value at Visit | 0.44 (0.020)
  Change From BL at Day 2 | 0.01 (0.032)
  Change From BL at Day 4 | 0.01 (0.024)
  Change From BL at Day 8 | 0.00 (0.023)
  Change From BL at Day 15 | 0.00 (0.018)
  Change From BL at Day 29 | -0.01 (0.019)
  Change From BL at Day 43 | 0.00 (0.025)
  Change From BL at Day 57 | -0.01 (0.027)
  Change From BL at Day 71 | 0.00 (0.027)
  Change From BL at Day 85 | 0.00 (0.029)
  Change From BL at Day 113 | 0.01 (0.029)
  Post-BL Minimum Change From BL | -0.02 (0.020)
  Post-BL Maximum Change From BL | 0.02 (0.022)

42. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Hemoglobin Concentration
Description: as for outcome 36
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: gram per Liter (g/L)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
gram per Liter (g/L)
  Baseline (BL) - Value at Visit | 149.38 (8.065)
  Change From BL at Day 2 | 3.94 (10.056)
  Change From BL at Day 4 | 5.38 (7.571)
  Change From BL at Day 8 | 0.88 (6.551)
  Change From BL at Day 15 | -2.50 (6.439)
  Change From BL at Day 29 | -2.50 (7.062)
  Change From BL at Day 43 | -0.56 (6.345)
  Change From BL at Day 57 | -1.94 (8.330)
  Change From BL at Day 71 | 0.94 (7.505)
  Change From BL at Day 85 | 0.88 (7.881)
  Change From BL at Day 113 | 3.19 (9.086)
  Post-BL Minimum Change From BL | -8.13 (6.076)
  Post-BL Maximum Change From BL | 9.63 (5.608)

43. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Lymphocytes, Absolute Count
Description: as for outcome 36
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: *10^9 cells per Liter
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
*10^9 cells per Liter
  Baseline (BL) - Value at Visit | 1.65 (0.691)
  Change From BL at Day 2 | 0.10 (0.381)
  Change From BL at Day 4 | 0.37 (0.780)
  Change From BL at Day 8 | 0.04 (0.595)
  Change From BL at Day 15 | -0.09 (0.599)
  Change From BL at Day 29 | -0.01 (0.422)
  Change From BL at Day 43 | 0.07 (0.470)
  Change From BL at Day 57 | 0.01 (0.464)
  Change From BL at Day 71 | 0.06 (0.372)
  Change From BL at Day 85 | 0.02 (0.397)
  Change From BL at Day 113 | 0.04 (0.585)
  Post-BL Minimum Change From BL | -0.35 (0.447)
  Post-BL Maximum Change From BL | 0.61 (0.633)

44. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Monocytes, Absolute Count
Description: as for outcome 36
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: *10^9 cells per Liter
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
*10^9 cells per Liter
  Baseline (BL) - Value at Visit | 0.35 (0.087)
  Change From BL at Day 2 | -0.04 (0.098)
  Change From BL at Day 4 | -0.03 (0.111)
  Change From BL at Day 8 | -0.04 (0.100)
  Change From BL at Day 15 | -0.01 (0.136)
  Change From BL at Day 29 | -0.01 (0.112)
  Change From BL at Day 43 | -0.03 (0.082)
  Change From BL at Day 57 | -0.04 (0.091)
  Change From BL at Day 71 | -0.03 (0.075)
  Change From BL at Day 85 | -0.04 (0.096)
  Change From BL at Day 113 | -0.02 (0.112)
  Post-BL Minimum Change From BL | -0.10 (0.080)
  Post-BL Maximum Change From BL | 0.11 (0.112)

45. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Total Neutrophils, Absolute Count
Description: as for outcome 36
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: *10^9 cells per Liter
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
*10^9 cells per Liter
  Baseline (BL) - Value at Visit | 3.57 (0.869)
  Change From BL at Day 2 | -0.24 (0.959)
  Change From BL at Day 4 | 0.12 (0.950)
  Change From BL at Day 8 | -0.19 (0.809)
  Change From BL at Day 15 | 0.19 (1.043)
  Change From BL at Day 29 | 0.23 (1.063)
  Change From BL at Day 43 | 0.06 (0.961)
  Change From BL at Day 57 | -0.24 (0.758)
  Change From BL at Day 71 | -0.06 (0.824)
  Change From BL at Day 85 | -0.31 (0.686)
  Change From BL at Day 113 | -0.27 (0.695)
  Post-BL Minimum Change From BL | -0.86 (0.708)
  Post-BL Maximum Change From BL | 1.16 (0.968)

46. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Platelet Count
Description: as for outcome 36
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: *10^9 cells per Liter
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
*10^9 cells per Liter
  Baseline (BL) - Value at Visit | 231.50 (47.880)
  Change From BL at Day 2 | -2.13 (25.469)
  Change From BL at Day 4 | -3.69 (22.330)
  Change From BL at Day 8 | 0.06 (20.612)
  Change From BL at Day 15 | 7.25 (23.023)
  Change From BL at Day 29 | 12.50 (26.967)
  Change From BL at Day 43 | 9.88 (30.265)
  Change From BL at Day 57 | 10.94 (18.908)
  Change From BL at Day 71 | 5.50 (34.131)
  Change From BL at Day 85 | 0.50 (30.542)
  Change From BL at Day 113 | 2.94 (23.778)
  Post-BL Minimum Change From BL | -27.31 (17.984)
  Post-BL Maximum Change From BL | 36.50 (26.473)

47. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: Red Blood Cell Count
Description: as for outcome 36
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: *10^12 cells per Liter
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
*10^12 cells per Liter
  Baseline (BL) - Value at Visit | 4.86 (0.304)
  Change From BL at Day 2 | 0.09 (0.327)
  Change From BL at Day 4 | 0.16 (0.247)
  Change From BL at Day 8 | -0.02 (0.235)
  Change From BL at Day 15 | -0.07 (0.196)
  Change From BL at Day 29 | -0.09 (0.209)
  Change From BL at Day 43 | -0.09 (0.226)
  Change From BL at Day 57 | -0.11 (0.289)
  Change From BL at Day 71 | -0.04 (0.266)
  Change From BL at Day 85 | -0.04 (0.334)
  Change From BL at Day 113 | 0.02 (0.337)
  Post-BL Minimum Change From BL | -0.31 (0.242)
  Post-BL Maximum Change From BL | 0.26 (0.213)

48. Secondary Outcome: Change From Baseline in Hematology Laboratory Test Results by Timepoint: White Blood Cell Count
Description: as for outcome 36
Time Frame: Baseline and Days 2, 4, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: *10^9 cells per Liter
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
*10^9 cells per Liter
  Baseline (BL) - Value at Visit | 5.74 (1.565)
  Change From BL at Day 2 | -0.17 (1.213)
  Change From BL at Day 4 | 0.33 (1.285)
  Change From BL at Day 8 | -0.20 (1.222)
  Change From BL at Day 15 | 0.09 (1.400)
  Change From BL at Day 29 | 0.21 (1.026)
  Change From BL at Day 43 | 0.11 (1.162)
  Change From BL at Day 57 | -0.27 (1.125)
  Change From BL at Day 71 | -0.01 (1.006)
  Change From BL at Day 85 | -0.34 (1.064)
  Change From BL at Day 113 | -0.24 (1.332)
  Post-BL Minimum Change From BL | -1.07 (1.071)
  Post-BL Maximum Change From BL | 1.29 (0.997)

49. Secondary Outcome: Number of Participants by Test Results for Blood in Urine by Timepoint
Description: Urine samples were collected from participants at the indicated timepoints for evaluation of urinalysis parameters. The number of participants with test results for blood in urine of 0 (Absent), +1 (Trace), +2 (Positive), and +3/+4 (Strong Positive) at baseline and each timepoint are reported. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 8, 29, 57, 85, and 113
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
Participants
  Baseline: 0 (Absent) | 15
  Baseline: +1 (Trace) | 1
  Baseline: +2 (Positive) | 0
  Baseline: +3/+4 (Strong Positive) | 0
  Day 2: 0 (Absent) | 16
  Day 2: +1 (Trace) | 0
  Day 2: +2 (Positive) | 0
  Day 2: +3/+4 (Strong Positive) | 0
  Day 8: 0 (Absent) | 15
  Day 8: +1 (Trace) | 1
  Day 8: +2 (Positive) | 0
  Day 8: +3/+4 (Strong Positive) | 0
  Day 29: 0 (Absent) | 16
  Day 29: +1 (Trace) | 0
  Day 29: +2 (Positive) | 0
  Day 29: +3/+4 (Strong Positive) | 0
  Day 57: 0 (Absent) | 16
  Day 57: +1 (Trace) | 0
  Day 57: +2 (Positive) | 0
  Day 57: +3/+4 (Strong Positive) | 0
  Day 85: 0 (Absent) | 16
  Day 85: +1 (Trace) | 0
  Day 85: +2 (Positive) | 0
  Day 85: +3/+4 (Strong Positive) | 0
  Day 113: 0 (Absent) | 15
  Day 113: +1 (Trace) | 1
  Day 113: +2 (Positive) | 0
  Day 113: +3/+4 (Strong Positive) | 0

50. Secondary Outcome: Number of Participants by Test Results for Glucose in Urine by Timepoint
Description: Urine samples were collected from participants at the indicated timepoints for evaluation of urinalysis parameters. The number of participants with test results for glucose in urine of 0 (Absent), +1 (Trace), +2 (Positive), and +3/+4 (Strong Positive) at baseline and each timepoint are reported. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 8, 29, 57, 85, and 113
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
Participants
  Baseline: 0 (Absent) | 16
  Baseline: +1 (Trace) | 0
  Baseline: +2 (Positive) | 0
  Baseline: +3/+4 (Strong Positive) | 0
  Day 2: 0 (Absent) | 16
  Day 2: +1 (Trace) | 0
  Day 2: +2 (Positive) | 0
  Day 2: +3/+4 (Strong Positive) | 0
  Day 8: 0 (Absent) | 16
  Day 8: +1 (Trace) | 0
  Day 8: +2 (Positive) | 0
  Day 8: +3/+4 (Strong Positive) | 0
  Day 29: 0 (Absent) | 16
  Day 29: +1 (Trace) | 0
  Day 29: +2 (Positive) | 0
  Day 29: +3/+4 (Strong Positive) | 0
  Day 57: 0 (Absent) | 16
  Day 57: +1 (Trace) | 0
  Day 57: +2 (Positive) | 0
  Day 57: +3/+4 (Strong Positive) | 0
  Day 85: 0 (Absent) | 16
  Day 85: +1 (Trace) | 0
  Day 85: +2 (Positive) | 0
  Day 85: +3/+4 (Strong Positive) | 0
  Day 113: 0 (Absent) | 15
  Day 113: +1 (Trace) | 1
  Day 113: +2 (Positive) | 0
  Day 113: +3/+4 (Strong Positive) | 0

51. Secondary Outcome: Number of Participants by Test Results for Protein in Urine by Timepoint
Description: Urine samples were collected from participants at the indicated timepoints for evaluation of urinalysis parameters. The number of participants with test results for protein in urine of 0 (Absent), +1 (Trace), +2 (Positive), and +3/+4 (Strong Positive) at baseline and each timepoint are reported. Baseline was defined as the participant's last sample prior to initiation of study drug.
Time Frame: Baseline and Days 2, 8, 29, 57, 85, and 113
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
Participants
  Baseline: 0 (Absent) | 16
  Baseline: +1 (Trace) | 0
  Baseline: +2 (Positive) | 0
  Baseline: +3/+4 (Strong Positive) | 0
  Day 2: 0 (Absent) | 16
  Day 2: +1 (Trace) | 0
  Day 2: +2 (Positive) | 0
  Day 2: +3/+4 (Strong Positive) | 0
  Day 8: 0 (Absent) | 16
  Day 8: +1 (Trace) | 0
  Day 8: +2 (Positive) | 0
  Day 8: +3/+4 (Strong Positive) | 0
  Day 29: 0 (Absent) | 16
  Day 29: +1 (Trace) | 0
  Day 29: +2 (Positive) | 0
  Day 29: +3/+4 (Strong Positive) | 0
  Day 57: 0 (Absent) | 15
  Day 57: +1 (Trace) | 1
  Day 57: +2 (Positive) | 0
  Day 57: +3/+4 (Strong Positive) | 0
  Day 85: 0 (Absent) | 15
  Day 85: +1 (Trace) | 1
  Day 85: +2 (Positive) | 0
  Day 85: +3/+4 (Strong Positive) | 0
  Day 113: 0 (Absent) | 16
  Day 113: +1 (Trace) | 0
  Day 113: +2 (Positive) | 0
  Day 113: +3/+4 (Strong Positive) | 0

52. Secondary Outcome: Change From Baseline in Vital Signs by Timepoint: Diastolic Blood Pressure
Description: Vital signs were measured prior to blood sampling while the participant was in a supine position after they had been resting for at least 5 minutes. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last value prior to initiation of study drug.
Time Frame: Baseline and Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millimeters of mercury (mmHg)
  Baseline (BL) - Value at Visit | 66.1 (5.77)
  Change From BL at Day 2 | -0.8 (4.99)
  Change From BL at Day 4 | 2.4 (5.21)
  Change From BL at Day 6 | 3.2 (5.43)
  Change From BL at Day 8 | 2.7 (5.41)
  Change From BL at Day 11 | 1.4 (5.11)
  Change From BL at Day 15 | 1.7 (4.24)
  Change From BL at Day 22 | 3.2 (5.46)
  Change From BL at Day 29 | 2.6 (5.67)
  Change From BL at Day 36 | 1.3 (4.48)
  Change From BL at Day 43 | 1.0 (5.18)
  Change From BL at Day 50 | 3.4 (6.49)
  Change From BL at Day 57 | -0.3 (4.64)
  Change From BL at Day 71 | 1.1 (5.50)
  Change From BL at Day 85 | 1.3 (4.52)
  Change From BL at Day 113 | 1.3 (4.73)
  Post-BL Minimum Change From BL | -5.2 (3.08)
  Post-BL Maximum Change From BL | 8.1 (4.39)

53. Secondary Outcome: Change From Baseline in Vital Signs by Timepoint: Pulse Rate
Description: as for outcome 52
Time Frame: Baseline and Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
beats per minute
  Baseline (BL) - Value at Visit | 61.3 (7.25)
  Change From BL at Day 2 | -0.6 (4.72)
  Change From BL at Day 4 | 1.3 (4.90)
  Change From BL at Day 6 | 5.8 (7.06)
  Change From BL at Day 8 | 7.7 (8.58)
  Change From BL at Day 11 | 9.9 (10.41)
  Change From BL at Day 15 | 6.9 (5.71)
  Change From BL at Day 22 | 10.2 (9.22)
  Change From BL at Day 29 | 8.4 (9.24)
  Change From BL at Day 36 | 6.3 (7.59)
  Change From BL at Day 43 | 6.2 (7.93)
  Change From BL at Day 50 | 10.4 (6.98)
  Change From BL at Day 57 | 7.5 (6.75)
  Change From BL at Day 71 | 4.7 (7.07)
  Change From BL at Day 85 | 6.9 (9.48)
  Change From BL at Day 113 | 7.4 (8.16)
  Post-BL Minimum Change From BL | -3.1 (4.46)
  Post-BL Maximum Change From BL | 18.1 (6.29)

54. Secondary Outcome: Change From Baseline in Vital Signs by Timepoint: Respiratory Rate
Description: as for outcome 52
Time Frame: Baseline and Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
breaths per minute
  Baseline (BL) - Value at Visit | 15.5 (1.51)
  Change From BL at Day 2 | 0.6 (1.50)
  Change From BL at Day 4 | 0.3 (1.89)
  Change From BL at Day 6 | -0.5 (2.00)
  Change From BL at Day 8 | 0.8 (2.64)
  Change From BL at Day 11 | 0.1 (2.55)
  Change From BL at Day 15 | -0.1 (2.38)
  Change From BL at Day 22 | -0.1 (2.60)
  Change From BL at Day 29 | 0.2 (2.10)
  Change From BL at Day 36 | 0.9 (1.54)
  Change From BL at Day 43 | -0.3 (1.88)
  Change From BL at Day 50 | 0.3 (2.32)
  Change From BL at Day 57 | 0.2 (2.14)
  Change From BL at Day 71 | -0.3 (2.02)
  Change From BL at Day 85 | -0.4 (2.33)
  Change From BL at Day 113 | 0.4 (2.47)
  Post-BL Minimum Change From BL | -3.0 (1.83)
  Post-BL Maximum Change From BL | 2.7 (1.82)

55. Secondary Outcome: Change From Baseline in Vital Signs by Timepoint: Systolic Blood Pressure
Description: as for outcome 52
Time Frame: Baseline and Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millimeters of mercury (mmHg)
  Baseline (BL) - Value at Visit | 106.8 (7.26)
  Change From BL at Day 2 | -1.6 (6.49)
  Change From BL at Day 4 | 2.4 (5.82)
  Change From BL at Day 6 | 3.6 (5.86)
  Change From BL at Day 8 | 3.5 (8.16)
  Change From BL at Day 11 | 5.1 (8.05)
  Change From BL at Day 15 | 2.5 (4.97)
  Change From BL at Day 22 | 4.8 (7.46)
  Change From BL at Day 29 | 3.2 (8.84)
  Change From BL at Day 36 | 2.2 (7.49)
  Change From BL at Day 43 | 2.0 (5.97)
  Change From BL at Day 50 | 5.2 (8.95)
  Change From BL at Day 57 | 2.2 (7.19)
  Change From BL at Day 71 | 1.2 (6.35)
  Change From BL at Day 85 | 2.0 (8.68)
  Change From BL at Day 113 | 1.1 (8.75)
  Post-BL Minimum Change From BL | -4.6 (5.76)
  Post-BL Maximum Change From BL | 10.9 (7.47)

56. Secondary Outcome: Change From Baseline in Vital Signs by Timepoint: Temperature (Axillary)
Description: as for outcome 52
Time Frame: Baseline and Days 2, 4, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: degrees Celsius (C)
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
degrees Celsius (C)
  Baseline (BL) - Value at Visit | 36.20 (0.239)
  Change From BL at Day 2 | -0.12 (0.281)
  Change From BL at Day 4 | 0.01 (0.263)
  Change From BL at Day 6 | -0.09 (0.532)
  Change From BL at Day 8 | -0.08 (0.217)
  Change From BL at Day 11 | -0.18 (0.414)
  Change From BL at Day 15 | -0.06 (0.515)
  Change From BL at Day 22 | -0.14 (0.352)
  Change From BL at Day 29 | -0.11 (0.433)
  Change From BL at Day 36 | -0.19 (0.313)
  Change From BL at Day 43 | -0.16 (0.318)
  Change From BL at Day 50 | -0.16 (0.418)
  Change From BL at Day 57 | 0.02 (0.382)
  Change From BL at Day 71 | -0.09 (0.360)
  Change From BL at Day 85 | -0.21 (0.260)
  Change From BL at Day 113 | -0.02 (0.297)
  Post-BL Minimum Change From BL | -0.61 (0.260)
  Post-BL Maximum Change From BL | 0.43 (0.357)

57. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Results by Timepoint: Heart Rate
Description: The 12-lead electrocardiogram (ECG) measurements were collected in triplicate (three consecutive interpretable ECGs within 5 minutes) after the participant had been in a supine position for at least 10 minutes. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit, including repeat and unscheduled tests. Baseline was defined as the participant's last value prior to initiation of study drug.
Time Frame: Baseline and Days 2, 4, 6, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
beats per minute
  Baseline (BL) - Value at Visit | 59.90 (5.588)
  Change From BL at Day 2 | -0.67 (3.656)
  Change From BL at Day 4 | 2.50 (3.978)
  Change From BL at Day 6 | 6.52 (6.491)
  Change From BL at Day 8 | 8.63 (7.574)
  Change From BL at Day 15 | 6.58 (4.250)
  Change From BL at Day 29 | 8.10 (8.675)
  Change From BL at Day 43 | 6.96 (7.946)
  Change From BL at Day 57 | 6.42 (5.793)
  Change From BL at Day 71 | 5.42 (6.976)
  Change From BL at Day 85 | 8.25 (8.234)
  Change From BL at Day 113 | 7.15 (6.442)
  Post-BL Minimum Change From BL | -2.21 (2.638)
  Post-BL Maximum Change From BL | 15.52 (6.259)

58. Secondary Outcome: Change From Baseline in ECG Results by Timepoint: PR Duration
Description: as for outcome 57
Time Frame: Baseline and Days 2, 4, 6, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millisecond
  Baseline (BL) - Value at Visit | 160.21 (16.023)
  Change From BL at Day 2 | 0.81 (12.767)
  Change From BL at Day 4 | -0.10 (9.229)
  Change From BL at Day 6 | -1.90 (9.998)
  Change From BL at Day 8 | -4.13 (12.692)
  Change From BL at Day 15 | -1.73 (14.577)
  Change From BL at Day 29 | -4.10 (10.197)
  Change From BL at Day 43 | -1.79 (13.850)
  Change From BL at Day 57 | -1.52 (10.352)
  Change From BL at Day 71 | -1.29 (9.008)
  Change From BL at Day 85 | -5.02 (12.450)
  Change From BL at Day 113 | -1.52 (6.576)
  Post-BL Minimum Change From BL | -15.21 (11.517)
  Post-BL Maximum Change From BL | 8.83 (9.000)

59. Secondary Outcome: Change From Baseline in ECG Results by Timepoint: QRS Duration
Description: as for outcome 57
Time Frame: Baseline and Days 2, 4, 6, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millisecond
  Baseline (BL) - Value at Visit | 98.15 (9.074)
  Change From BL at Day 2 | 0.75 (5.514)
  Change From BL at Day 4 | 1.40 (3.077)
  Change From BL at Day 6 | -0.71 (3.052)
  Change From BL at Day 8 | -0.48 (4.169)
  Change From BL at Day 15 | -0.40 (3.221)
  Change From BL at Day 29 | -1.00 (5.594)
  Change From BL at Day 43 | -0.65 (2.327)
  Change From BL at Day 57 | -1.54 (2.494)
  Change From BL at Day 71 | 0.77 (3.429)
  Change From BL at Day 85 | -0.46 (3.494)
  Change From BL at Day 113 | -0.92 (3.782)
  Post-BL Minimum Change From BL | -4.19 (3.592)
  Post-BL Maximum Change From BL | 4.50 (3.475)

60. Secondary Outcome: Change From Baseline in ECG Results by Timepoint: QT Duration
Description: as for outcome 57
Time Frame: Baseline and Days 2, 4, 6, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millisecond
  Baseline (BL) - Value at Visit | 398.31 (27.123)
  Change From BL at Day 2 | -1.35 (11.351)
  Change From BL at Day 4 | -10.00 (13.856)
  Change From BL at Day 6 | -12.31 (19.791)
  Change From BL at Day 8 | -15.69 (15.037)
  Change From BL at Day 15 | -9.90 (13.857)
  Change From BL at Day 29 | -11.83 (19.322)
  Change From BL at Day 43 | -11.96 (13.863)
  Change From BL at Day 57 | -7.56 (16.498)
  Change From BL at Day 71 | -4.94 (19.933)
  Change From BL at Day 85 | -9.75 (23.282)
  Change From BL at Day 113 | -9.21 (20.349)
  Post-BL Minimum Change From BL | -30.35 (14.706)
  Post-BL Maximum Change From BL | 9.60 (12.064)

61. Secondary Outcome: Change From Baseline in ECG Results by Timepoint: QTcB Duration (Bazett's Correction Formula)
Description: as for outcome 57
Time Frame: Baseline and Days 2, 4, 6, 8, 15, 29, 43, 57, 71, 85, and 113
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millisecond
  Baseline (BL) - Value at Visit | 398.04 (19.275)
  Change From BL at Day 2 | -3.81 (10.367)
  Change From BL at Day 4 | -2.29 (8.759)
  Change From BL at Day 6 | 7.33 (8.549)
  Change From BL at Day 8 | 10.08 (13.968)
  Change From BL at Day 15 | 10.50 (10.870)
  Change From BL at Day 29 | 12.69 (12.031)
  Change From BL at Day 43 | 8.81 (13.699)
  Change From BL at Day 57 | 12.00 (9.509)
  Change From BL at Day 71 | 12.25 (12.194)
  Change From BL at Day 85 | 15.27 (13.029)
  Change From BL at Day 113 | 12.08 (13.229)
  Post-BL Minimum Change From BL | -7.27 (8.817)
  Post-BL Maximum Change From BL | 24.23 (11.165)

62. Secondary Outcome: Change From Baseline in ECG Results by Timepoint: QTcF Duration (Fridericia's Correction Formula)
Description: as for outcome 57
Time Frame: Baseline and Days 2, 4, 6, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millisecond
  Baseline (BL) - Value at Visit | 397.90 (20.554)
  Change From BL at Day 2 | -2.98 (8.968)
  Change From BL at Day 4 | -4.94 (9.038)
  Change From BL at Day 6 | 1.21 (9.739)
  Change From BL at Day 8 | 1.31 (9.708)
  Change From BL at Day 15 | 3.56 (10.109)
  Change From BL at Day 29 | 4.33 (8.384)
  Change From BL at Day 43 | 1.69 (8.274)
  Change From BL at Day 57 | 5.31 (8.893)
  Change From BL at Day 71 | 6.40 (11.109)
  Change From BL at Day 85 | 6.71 (12.243)
  Change From BL at Day 113 | 4.81 (12.931)
  Post-BL Minimum Change From BL | -8.21 (8.174)
  Post-BL Maximum Change From BL | 14.77 (10.366)

63. Secondary Outcome: Change From Baseline in ECG Results by Timepoint: RR Duration
Description: as for outcome 57
Time Frame: Baseline and Days 2, 4, 6, 8, 15, 29, 43, 57, 71, 85, and 113
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
millisecond
  Baseline (BL) - Value at Visit | 1001.06 (93.082)
  Change From BL at Day 2 | 12.73 (66.160)
  Change From BL at Day 4 | -36.04 (60.573)
  Change From BL at Day 6 | -94.79 (99.788)
  Change From BL at Day 8 | -119.67 (106.349)
  Change From BL at Day 15 | -96.56 (67.805)
  Change From BL at Day 29 | -114.08 (126.347)
  Change From BL at Day 43 | -97.98 (109.011)
  Change From BL at Day 57 | -92.98 (87.990)
  Change From BL at Day 71 | -82.29 (112.001)
  Change From BL at Day 85 | -115.87 (122.073)
  Change From BL at Day 113 | -101.02 (98.269)
  Post-BL Minimum Change From BL | -205.40 (91.026)
  Post-BL Maximum Change From BL | 40.25 (49.296)

64. Secondary Outcome: Number of Participants With Concomitant Medications
Description: The original terms recorded by the investigator for concomitant medications were standardized by the sponsor by assigning preferred terms. The duration of treatment with the concomitant medications ranged from 1 day to 5 days. Except for 1 participant who was treated during the in-clinic period (Days -1 to 4), all other concomitant medications were recorded during the ambulatory period (Days 6 to 113).
Time Frame: From screening to study completion (20 weeks)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab
Number analyzed (Participants) | 16
Participants
  Total Participants with at Least 1 Treatment | 6
  Analgesics - Paracetamol | 1
  Antitrichomonal Agents - Tinidazole | 1
  Cephalosporin Antibiotics - Cefadroxil | 1
  Cephalosporin Antibiotics - Cefminox | 1
  Herbal, Homeopathic, and Dietary Supplements | 1
  Non-Steroidal Anti-Inflammatories - Pranoprofen | 1
  Proton Pump Inhibitors - Pantoprazole | 1
  Salicylates - Aspirin DL-Lysine | 1
  Supplements - Potassium Chloride | 1
  Supplements - Sodium Chloride | 1
  Vitamins and Minerals - Ascorbic Acid | 1

ADVERSE EVENTS:
Time Frame: From screening to study completion (20 weeks)
Description: Investigators sought information on adverse events (AEs) at each contact with participants. After informed consent but prior to initiation of study drug, only serious AEs (SAEs) caused by a protocol-mandated intervention were to be reported. After initiation of study drug, all AEs, regardless of relationship to study drug, were to be reported until the participant completed his last study visit. After this period, any SAEs believed to be related to prior study drug treatment were to be reported.
Arm/Group | Emicizumab
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 14/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Emicizumab (N=16)
Leukopenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Conjunctivitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pericoronitis (Infections and infestations) | 1
Injury (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Blood creatinine phosphokinase increased (Investigations) | 4
C-reactive protein increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT03380780/Prot_SAP_000.pdf